CLINICAL TRIAL: NCT01411488
Title: Randomized Controlled Study of the Effects of Two Fecal Management Systems on Incidence of Anal Erosion.
Brief Title: Comparative Study Between Two Fecal Management Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Bard Ltd (Industry)
Responsible Party: Principal Investigator, Nancy M. Albert, Ph.D., Cleveland Clinic Foundation, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-1098
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Anal Erosion
Keywords: Focus: anal erosion

STUDY DESIGN:
Intervention Model Description: 2 Groups were randomly assigned to 1 of 2 different fecal management systems
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal Management System- Company 1 (Experimental): 80 adult patients to be randomly assigned to receive a fecal management system by Bard Medical
  Interventions: Device: Fecal management system
- Fecal Management System- Company 2 (Active Comparator): 80 adult patients to be randomly assigned to receive a fecal management system by ConvaTec
  Interventions: Device: Fecal management system

INTERVENTIONS:
Device: Fecal management system — rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions

SUMMARY:
The purpose of the study is to determine the prevalence of anal erosions within a 14 day period among adult ICU patients at Cleveland Clinic Main Campus who receive one of two fecal management systems (FMS).

Null Hypothesis: There is no difference in the rates of anal erosion between the twp fecal management systems in a 14 day period.

Alternative Hypothesis: One fecal management system is no worse than the second fecal management system in the development of anal erosion.

DETAILED DESCRIPTION:
PURPOSE: To compare the incidence of anal erosion between 2 indwelling fecal management systems. Anal erosion was defi ned as localized mucous membrane tissue impairments of the anal canal caused by corrosive fecal enzymes and/or indwelling devices. DESIGN: Randomized comparative effectiveness clinical trial comparing 2 commercially available indwelling fecal management systems. SUBJECTS AND SETTING: The target population was adults cared for on medical, surgical, and neurological intensive care units (ICUs) and non-ICU units with an order for indwelling fecal management system placement. The research setting was a 1200-bed quaternary-care medical center in the Midwestern United States. 90 patients were enrolled in the study. The number who started and completed the study; 41 of 47 received system A and 38 of 43 received system B. Subjects' mean age was 64 ± 13.6 years (mean ± SD), and 52% were female.

ELIGIBILITY:
Inclusion Criteria:

* Bedfast patients who need to have liquid or semi-liquid stool contained away from the body to prevent skin breakdown or contamination of existing wounds

  * Liquid to semi-liquid stool incontinence for past three days that is expected to last for extended period due to poor response to anti-diarrheal treatment
  * Absence of contraindications listed in Exclusion Criteria
  * If on subcutaneous anti-coagulation to prevent deep vein thrombosis, then can be included in study

Exclusion Criteria:

* Allergic to product components

  * Rectal or anal injury or active bleeding
  * Severe rectal or anal stricture or stenosis (distal rectum cannot accommodate the balloon), diseases of the rectal mucosa (i.e. severe proctitis, ischemic proctitis, mucosal lacerations)
  * Rectal or anal tumors
  * Severe hemorrhoids
  * Fecal impaction
  * Loss of rectal tone or prolapsed anal sphincter
  * History of Ileo-anal anastamosis or internal rectal pouch (e.g. S or J pouch)
  * Large Bowel (Colon) surgery or rectal surgery within the last year
  * Currently on heparin drip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Albert, PhD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An interim analysis was planned one 70+ patients completed data collection to determine futility vs continued recruitment, enrollment and data collection.
  The analysis presented represents the interim analysis as it was determines that we should stop further recruitment and enrollment based on study findings.
Pre-assignment Details: An interim analysis was completed; see recruitment details
Groups:
- Fecal Management System- Company 1: 47 adult patients to be randomly assigned to receive a fecal management system by Bard Medical
  Fecal management system: rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions
  Note, not all patients were retained
- Fecal Management System- Company 2: 43 adult patients to be randomly assigned to receive a fecal management system by ConvaTec
  Fecal management system: rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions
  Note: not all patients were retained
Period: Overall Study
Arm/Group | Fecal Management System- Company 1 | Fecal Management System- Company 2
Started | 41 | 38
Completed | 41 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fecal Management System- Company 1: 41 adult patients to be randomly assigned to receive a fecal management system by Bard Medical
  Fecal management system: rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions
  55% male; 60% had history of hemorrhoids
- Fecal Management System- Company 2: 38 adult patients to be randomly assigned to receive a fecal management system by ConvaTec
  Fecal management system: rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions
  45% male; 39.1% had history of hemorrhoids
- Total: Total of all reporting groups
Arm/Group | Fecal Management System- Company 1 | Fecal Management System- Company 2 | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (15.0) | 64.7 (12.3) | 64.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Anal Erosion Within 14 Days After Insertion of FMS
Description: anal erosion within 14 days after insertion of FMS
Time Frame: up to 14 days
Population: Pearson's chi square test (categorical data) and Wilcoxon test (continuous measures). Logistic regression was used to assess primary endpoint by time the device was in use.
Measure: Count of Participants; unit: Participants
Groups:
- Fecal Management System- Company 1: 41 adult patients to be randomly assigned to receive a fecal management system by Bard Medical
  Fecal management system: rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions
- Fecal Management System- Company 2: 38 adult patients to be randomly assigned to receive a fecal management system by ConvaTec
  Fecal management system: rectal tubes/fecal management systems: we compared products to determine if there is a difference in the incidence of anal erosions
Arm/Group | Fecal Management System- Company 1 | Fecal Management System- Company 2
Number analyzed (Participants) | 41 | 38
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: During data collection for each subject. No follow up data collection
Description: Since rectal tube insertion is usual care, patient adverse evens were not recorded, only adverse events related to rectal tube care specifically
Arm/Group | Fecal Management System- Company 1 | Fecal Management System- Company 2
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38
Other Adverse Events (participants affected / at risk) | 3/41 | 2/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Management System- Company 1 (N=41) | Fecal Management System- Company 2 (N=38)
did not get to day 1 or could not tolerate (Gastrointestinal disorders) | 3 (3) | 2 (2) — rectal tube was not maintained for 24 hours

LIMITATIONS AND CAVEATS:
Single center Small sample size restricted to medical intensive care and other adults requiring rectal tube placement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No